CLINICAL TRIAL: NCT02005796
Title: Bioavailability of Anthocyanins of Blue Potatoes as Compared With Bilberries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, PhD, University of Turku
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Siniset perunat
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Postprandial Glycemia
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blue-fleshed potato tubers (Experimental): Intervention: Steam cooked mashed potato tubers
  Interventions: Other: Dietary intervention
- Yellow-fleshed potato tubers (Experimental): Intervention: Steam cooked mashed potato tubers
  Interventions: Other: Dietary intervention
- Bilberries and potato starch (Experimental): Intervention: A gel boiled with bilberries and potato starch
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention

SUMMARY:
In this study, the postprandial glycemia and insulinemia caused by boiled potato with blue-fleshed or yellow-fleshed tubers, or a gel prepared with bilberries and potato starch, is studied in healthy males. Additionally, the appearance and metabolism of the flavonoids and their metabolites is studied in plasma and urine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Male
* No regular medication
* No participation in a drug trial or blood donation within 2 months
* Non-smoker
* Signs informed consent
* Body mass index 18.5-27 kg/m2
* Fasting plasma cholesterol < 5.5 mmol/l
* Fasting plasma triacylglycerols < 2.6 mmol/l
* Fasting plasma glucose 4-6 mmol/l
* blood pressure <140/80 mmHg
* hemoglobin>130 g/l
* Fasting plasma alanine amino transferase (ALAT) <60 U/l (normal liver function)
* Fasting plasma thyroid-stimulating hormone (TSH) 0.4 - 4.5 mU/l (normal thyroid function)
* Fasting plasma creatinine <118 µmol/l (normal kidney function)

Exclusion Criteria:

* Regular smoking
* Alcohol abuse
* Regular medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Plasma glucose concentration | 20min, 40min, 60min, 90min, 120min, 180min, 240min
Plasma insulin concentration | 20min, 40min, 60min, 90min, 120min, 180min, 240min

SECONDARY OUTCOMES:
Concentrations and quality of flavonoid color compounds or their metabolites in plasma and urine (HPLC-measurement) | 20min, 40min, 60min, 90min, 120min, 180min, 240min
Concentrations and quality of flavonoid color compounds or their metabolites in plasma and urine (NMR-measurement) | 20min, 40min, 60min, 90min, 120min, 180min, 240min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biochemistry, University of Turku, University of Turku, Turku, Finland